CLINICAL TRIAL: NCT02572102
Title: Impact of Energy Drinks and Panax Ginseng on Heart Rhythm in Healthy Volunteers
Brief Title: Impact of Energy Drinks and Panax Ginseng on Heart Rhythm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of the Pacific (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 15-119
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Electrical Alternation of Heart; Blood Pressure
Keywords: ECG; Blood Pressure; Energy Drinks; Panax Ginseng
MeSH Terms: interventions — Energy Drinks; Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Energy Drink (Experimental): Two 16 ounce containers of an Energy Drink
  Interventions: Dietary Supplement: Energy Drink
- Panax Ginseng (Active Comparator): 800 mg of Panax Ginseng in 70 mL of cherry syrup, 20 mL of lime juice, 410 mL of carbonated water
  Interventions: Dietary Supplement: Panax Ginseng
- Placebo (Placebo Comparator): 70 mL of cherry syrup, 20 mL of lime juice, 410 mL of carbonated water
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Energy Drink — Energy Drink, two 16oz containers consumed in 45 minutes
  Arms: Energy Drink
Dietary Supplement: Panax Ginseng — Panax Ginseng, lime juice, water and cherry flavoring
  Arms: Panax Ginseng
Other: Placebo — Lime juice, water and cherry flavoring
  Arms: Placebo

SUMMARY:
To assess the cardiac effects of an energy drink and Panax Ginseng in healthy volunteers.

DETAILED DESCRIPTION:
Energy drinks are composed of a variety of ingredients such as caffeine, taurine, and panax ginseng amongst others. The safety and efficacy of these ingredients individually and in combination need further exploration. This study is designed to assess the electrocardiographic and blood pressure effects of energy drinks and panax ginseng in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults 18-40 years old.

Exclusion Criteria:

* Baseline corrected QT (QTc) interval greater than 440 milliseconds,
* blood pressure at initial screening appointment greater than 140/90 mmHg,
* concurrent use of prescriptions or OTC medications taken on a daily basis,
* pregnant females,
* patients with any baseline ECG abnormalities.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
QTc interval changes | 5.5 hours over 3 visits
Systolic blood pressure changes | 5.5 hours over 3 visits

SECONDARY OUTCOMES:
QT interval changes | 5.5 hours over 3 visits
PR interval changes | 5.5 hours over 3 visits
QRS duration changes | 5.5 hours over 3 visits
Heart rate changes | 5.5 hours over 3 visits
Diastolic blood pressure changes | 5.5 hours over 3 visits